CLINICAL TRIAL: NCT06240013
Title: Acute Effects of Foam Rolling and Proprioceptive Neuromuscular Facilitation Stretching During Warm-Up on Muscle Flexibility, Strength and Pain Threshold in Amateur Athletes
Brief Title: Acute Effects of Foam Rolling and Proprioceptive Neuromuscular Facilitation Stretching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-20-683
Record Dates: First submitted 2024-01-12; First posted 2024-02-02 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Athletes
Keywords: Muscle Stretching Exercises; Pain Threshold; Range of Motion, Articular; Muscle Strength
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Training Program (Experimental): 5 minutes of light aerobic cycling, unilateral 2*60 sec on dominant leg - 2 min foam rolling training in total
  Interventions: Other: Foam Rolling
- Group 2 Training Program (Experimental): 5 minutes of light aerobic cycling, unilateral 4*30 seconds on the dominant leg - 2 minutes in total proprioceptive neuromuscular facilitation stretching training
  Interventions: Other: Proprioceptive Neuromuscular Facilitation Stretching

INTERVENTIONS:
Other: Foam Rolling — Participants will take a long sitting position on a solid and flat surface, positioning their arms back and transferring their body weight to their palms. The foam roller to be applied to the dominant side will be placed under the hamstrings and slowly moved back and forth from the ischial tuberosity to the popliteal fossa, applying pressure for 2 minutes.
  Arms: Group 1 Training Program
Other: Proprioceptive Neuromuscular Facilitation Stretching — A PNF stretching protocol will be implemented with each participant assuming a tall sitting position on a solid, flat surface with their knees extended as much as possible. At this moment, the participant will be asked to perform maximum isometric hamstring muscle contraction for 5 seconds, followed by 5 seconds of relaxation and 20 seconds of stretching.
  Arms: Group 2 Training Program

SUMMARY:
The hamstring muscle is one of the key elements in rehabilitation programs and sports activities that enable the restoration of optimal muscle length. Decreased flexibility in the hamstring muscle may disrupt the biomechanics of the waist and pelvis, leading to low back pain or musculoskeletal disorders.

This study aims to investigate the acute effects of foam rolling and proprioceptive neuromuscular facilitation stretching during warm-up on muscle flexibility, strength, and pain threshold in amateur athletes. According to our research, there is no study in this field in the literature.

H1: There is a difference between the acute effects of foam rolling exercise and PNF stretching exercise on muscle flexibility during warm-up in amateur athletes.

H2: There is a difference between the effects of foam rolling and PNF stretching exercises used as warm-up exercises on muscle strength.

H3: Foam rolling and PNF stretching exercises applied to the Hamstring muscle as a warm-up exercise make a difference in the pain threshold of the lumbar region and Hamstring muscle.

DETAILED DESCRIPTION:
Stretching techniques used in athletes are frequently and widely used due to many effects such as changing range of motion, comfortable movement maintenance, and removal. There is no consensus in the literature on which of the static, dynamic, and proprioceptive neuromuscular facilitation stretching techniques is most effective, as opposed to the types of stretching for flexibility. There is no clear benefit of different stretching techniques to muscle performance. Accordingly, in the literature, it is seen that proprioceptive neuromuscular facilitation stretching techniques show a greater increase in joint range of motion compared to other stretching techniques.

Recently, the use of foam rolling has become widely used in sports applications due to similar effects seen in stretching and the hypothesized presence of a curative effect on muscle performance. There is not enough research on the extent of foam rolling during warm-up exercises to increase flexibility and muscle strength.

The hamstring muscle is one of the key elements in harmonious programs and sports activities that ensure the restoration of optimal muscle length. The emergence of the output in the hamstring muscle may disrupt the biomechanics of the waist and pelvis, causing low back pain or musculoskeletal disorders.

This study aims to investigate the acute effects of foam rolling and proprioceptive neuromuscular facilitation stretching on muscle input, strength, and pain intensity during nutrition in amateur athletes.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* Being an amateur athlete

Exclusion Criteria:

* Hypermobility
* History of hamstring injury in the last 6 months
* Diagnosed orthopedic problems
* Surgery in the lower extremity or spine
* Back pain
* Presence of systemic or neurological disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Hamstring Flexibility | Pre-intervention and immediately after the intervention
  Hamstring flexibility (mm) will be evaluated with the sit-reach test. Baseline® Sit and Reach Flexibility Measurement device will be used for testing. Participants will sit on the floor with their lower extremities extended and together; Their backs and hips will be supported against the wall, and the soles of their feet will be placed on the edge of the device. Participants will then extend their arms forward, with both hands facing down and one hand on top of the other (always the same hand on top). Participants will then be asked to lie forward and slide their hands as far as possible on the measurement scale without bending their knees. Measurements will be repeated three times and the average value will be recorded.
Hamstring Muscle Strength | Pre-intervention and immediately after the intervention
  Strength measurement of the participants' Hamstring muscles will be made using a digital hand dynamometer (J Tech Commender Muscle Tester). Participants will be instructed to sit in a fairly upright position in a chair, with their arms crossed in front of their chest and their legs hanging over the edge, with their knees and hips flexed at 90°. For isometric knee flexion muscle measurement evaluation, the dynamometer will be placed in the sural triceps region (5 cm proximal to the lateral malleolus). Participants press the dynamometer as hard as possible for three seconds, while the assessor will provide resistance, preventing any movement to achieve an isometric contraction.
Pain Threshold | Pre-intervention and immediately after the intervention
  An algometer (Dolorimeter) will be used to objectively measure pain threshold and pain tolerance. The pain threshold value due to the pressure to be applied to the hamstring muscle and waist area will be measured using an electronic algometer (Algometer, Baseline FDK 10) while the athlete is in a prone position on the bed. The algometer will be applied vertically to the most painful point, increasing the pressure by 1kg/cm2 every three seconds until the patient feels pain. The pressure value that causes the feeling of pain will be determined as the pain threshold.

SECONDARY OUTCOMES:
Lower Extremity Muscle Strength | Pre-intervention and immediately after the intervention
  A vertical jump test will be performed to evaluate the participants' lower extremity muscle strength. The measurement has two stages; measuring reach height, measuring jump height.
  1. Measuring reach height: The athlete stands with his feet flat on the ground. He/she is asked to raise his/her arms up from the side of the body. The point his fingers reach is recorded.
  2. Measuring the jump height: The athlete is asked to move away from the wall. The starting position is with feet shoulder-width apart and knees extended. After the hips and knees are bent, the athlete is asked to jump. The athlete reaches the highest point he can reach with his hands. The length of this point is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Elif E Safran, asst. prof., Study Director — Acibadem University; Hayri E Yılmaz, Principal Investigator — Acibadem University; Birce B Çelik, Study Chair — Acibadem University; Mahmut E Bükülmez, Study Chair — Acibadem University; Eren Çekiç, Study Chair — Acibadem University
Locations (1):
- Acibadem University, Istanbul, None Selected, Turkey (Türkiye)